CLINICAL TRIAL: NCT00770731
Title: A Phase I Study of Temsirolimus, Topotecan, and Bortezomib in Patients With Advanced Malignancy
Brief Title: Study of Temsirolimus, Topotecan, and Bortezomib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0425
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Advanced Cancer
Keywords: Torisel; Temsirolimus; Hycamtin; Topotecan hydrochloride; Velcade; Bortezomib; FDG-PET Scans; 18F-Fluoro-2-Deoxyglucose Positron Emission Tomography
MeSH Terms: interventions — temsirolimus; Topotecan; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Torisel + Hycamtin + Velcade (Experimental): Torisel starting Dose 5 mg Intravenously over 30-60 minutes, Days 1, 8, and 15 of 21 Day Cycle.
  Hycamtin starting Dose 0.8 mg/m^2 Intravenously over 30-60 minutes on Days 1 and 8 of 21 Day Cycle.
  Velcade starting Dose 0.3 mg/m^2 Intravenously over 1 minute on Days 1, 4, 8, and 11 of 21 Day Cycle.
  Interventions: Drug: Torisel (Temsirolimus); Drug: Hycamtin (Topotecan); Drug: Velcade (Bortezomib)
- Expansion Group (Experimental): Torisel + Hycamtin + Velcade Expansion Group
  Addition of 10 participants at highest tolerated dose level
  Interventions: Drug: Torisel (Temsirolimus); Drug: Hycamtin (Topotecan); Drug: Velcade (Bortezomib)

INTERVENTIONS:
Drug: Torisel (Temsirolimus) — Starting Dose 5 mg Intravenously over 30-60 minutes, Days 1, 8, and 15 of 21 Day Cycle
  Other Names: Temsirolimus; CCI-779
Drug: Hycamtin (Topotecan) — Starting Dose 0.8 mg/m^2 Intravenously over 30-60 minutes on Days 1 and 8 of 21 Day Cycle
  Other Names: Topotecan; Topotecan Hydrochloride
Drug: Velcade (Bortezomib) — Starting Dose 0.3 mg/m^2 Intravenously over 1 minute on Days 1, 4, 8, and 11 of 21 Day Cycle
  Other Names: Bortezomib; LDP-341; MLN341; PS-341

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of Torisel (temsirolimus), Hycamtin (topotecan hydrochloride), and Velcade (bortezomib) that can be given, in combination, to patients with advanced cancer that has spread or is unable to be surgically removed. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Temsirolimus is designed to block pathways that control important events such as the growth of blood vessels that are vital for the growth of cancer. This may cause cancer cells to die.

Topotecan hydrochloride is designed to block the function of important proteins in cancer cells. These proteins, when active, allow a cell's genes to duplicate and for the cancer cells to divide.

Bortezomib is designed to block the function of important proteins in cancer cells. These proteins control the destruction of proteins in tumor cells, which is important for their growth. This may cause cancer cells to die.

Study Drug Dose Level:

If you are found to be eligible to take part in this study, you will be enrolled into a group of about 3-6 participants that are receiving the same drug combination. The first group of participants will receive the lowest dose of the drug combination. The next group of participants will receive the next highest dose of the drug combination. The third group will receive an even higher dose than that. This process will continue until the study doctor finds the highest safe dose of the drug combination. The dose that you receive will depend on when you are enrolled in this study and the safety data that is available at that time. The dose that you receive may be lowered if you do not tolerate the study drug combination well. You will not receive any doses of the study drug higher than the dose you are first assigned to.

Once the highest tolerated dose is found, up to 10 more participants will be added at that dose level. This is called an Expansion Group.

Study Drug Administration:

Temsirolimus, topotecan, and bortezomib will be given in "cycles." Cycles will be about 21 days long or longer, depending on any side effects you may experience.

On Days 1, 8, and 15 of each cycle, you will receive temsirolimus through a needle in your vein over about 30-60 minutes.

On Days 1 and 8 of each cycle, you will receive topotecan hydrochloride by vein over about 30-60 minutes.

On Days 1, 4, 8, and 11 of each cycle, you will receive bortezomib by vein over less than 1 minute.

While on study you will not be able to take any drugs that may interfere with the study drugs. You should talk with your doctor before taking any non-study drugs.

Study Visits:

Once a week during Cycle 1, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* If the doctor thinks it is needed, urine will be collected for routine tests.

If you are in the Expansion Group, then during Week 3 of Cycle 1, you will have a tumor biopsy to compare the activity of the tumor before treatment and after treatment has begun. This is done for research purposes only.

If you are in the Expansion Group, then 24-48 hours after starting Week 1 of Cycle 1, you will have a bone marrow aspiration performed. The tissue will be used to see how the study drug combination acts in the body and to learn the effect it may have on cancer cells. This is done for research purposes only.

During Week 1 of Cycle 2, you will have an ECG. After this, you will have extra ECGs if the doctor thinks it is needed.

During Week 1 of Cycles 2 and beyond, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* If the doctor thinks it is needed, urine may be collected for routine tests.

Once every 2 cycles (Cycles 2, 4, 6, and so on), you will have a CT or MRI scan to check the status of the disease.

FDG-PET Scans:

Every 2-3 months while you are on study and before Cycle 1 if you have not had a FDG-PET within the last 1 month, you may have a FDG-PET scan. You must fast for at least 6 hours before the FDG-PET scan. If you are a diabetic, you must fast for at least 4 hours before the FDG-PET scan. If it is needed, you may take drugs or drink water. The FDG-PET will be used to see if the activity of the cancers decreased with the drugs.

You will receive a small amount of FDG solution by vein. You will then rest in a quiet darkened room for 45-60 minutes before the PET scan. Pictures of your body will be taken using a PET scanner, which will about take 1 1/2 hours. The entire procedure should take about 3 hours.

Each time you have a FDG-PET scan, blood (either a finger stick or about 1 teaspoon) will be drawn to measure your blood sugar levels.

Length of Study Participation:

You will be on study for as long as you are benefiting. You will be taken off study if the disease gets worse or intolerable side effects occur.

End-of-Treatment Visit:

After you are off study, you will have an end-of-treatment visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests.

This is an investigational study. Temsirolimus, topotecan, and bortezomib are all FDA approved and commercially available. Temsirolimus is FDA approved for the treatment of renal cell cancer. Topotecan hydrochloride is FDA approved for the treatment of ovarian, small cell lung, and cervical cancers. Bortezomib is FDA approved for the treatment of multiple myeloma and mantle cell lymphoma. The use of these drugs together is investigational and authorized for use in research only.

Up to 80 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced or metastatic cancer that is refractory to standard therapy, relapsed after standard therapy, or have no standard therapy that improves survival by at least three months
2. Patients should be at least four weeks or 5 half lives from the last day of chemotherapy, and antibody or other biological therapy, whichever is shorter.
3. Patients should be at least four weeks from the last day of therapeutic radiation.
4. The Eastern Cooperative Oncology Group (ECOG) performance status </= 2 or Karnofsky >/= 60%.
5. Patients must have allowable organ and marrow function defined as: Absolute neutrophil count >/= 1,000/mL, Platelets >/=75,000/mL, Serum creatinine </= 2 * Upper Limit of Normal (ULN), Total bilirubin </= 2 * ULN, aminotransferase (ALT or SGPT) </= 3 * ULN, Fasting total cholesterol <= 350 mg/dL and triglyceride level <= 400 mg/dL.
6. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and will be advised to avoid pregnancy for 3 months after completion of therapy.
7. Ability to understand and the willingness to sign a written informed consent document.
8. Patients may not be receiving any other investigational agents and/or any other concurrent anticancer agents or therapies except for continuing on hormonal therapy in cases of prostate cancer.
9. Treatment on this study may begin within 24 hours after Phase 0 dose of temsirolimus.

Exclusion Criteria:

1. Patients with hemoptysis within 28 days prior to entering the study.
2. Patients with clinically significant unexplained bleeding within 28 days prior to entering the study.
3. Patients with clinically significant cardiovascular disease: • History of CVA within 6 months • Myocardial infarction or unstable angina within 6 months • Unstable angina pectoris
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics on Day 1.
5. Pregnant or lactating women.
6. History of hypersensitivity to bortezomib or any component of the bortezomib formulation.
7. History of hypersensitivity to topotecan or any component of the topotecan formulation.
8. History of hypersensitivity to temsirolimus or its metabolites (including sirolimus), polysorbate 80, or to any component of the formulation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of combination treatment with temsirolimus, topotecan, and bortezomib | 21 days
  MTD is defined as the highest dose in which the incidence of a dose limiting toxicity (DLT) is < 33%.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Karp, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org